CLINICAL TRIAL: NCT03260959
Title: Experience of the Father Following the Announcement of a First Pregnancy
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0073
Record Dates: First submitted 2017-08-22; First posted 2017-08-24 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2017-08

CONDITIONS: Family Relations; Behavior
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Father: Male having been the father of at least one pregnancy whatever the outcome (pregnancy pursued, or abortion)
  Interventions: Behavioral: Interview by hierarchical evocation's Method

INTERVENTIONS:
Behavioral: Interview by hierarchical evocation's Method — Interview to describe the experience of the man during the announcement of a pregnancy that it is expected or not.

SUMMARY:
Experience of the father following the announcement of a first pregnancy Its context, immediate reactions and actions. Possible impact of this moment of life a few months or years later?

ELIGIBILITY:
Inclusion Criteria:

- Male having been the father of at least one pregnancy whatever the outcome (pregnancy pursued, or abortion)

Exclusion Criteria:

* Patients with severe or neurological psychiatric disorders inducing significant cognitive impairment
* Patients who do not master the French language
* Patients who cannot give free and informed consent (guardianship, curatorship, safeguard of justice ...)

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Male having been the father of at least one pregnancy whatever the outcome (pregnancy pursued, or abortion)
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2017-11-10 (Actual)

PRIMARY OUTCOMES:
Interview by hierarchical evocation's method | 30-45 minutes
  Experience of the man during the announcement of a pregnancy that it is expected or not, without identification of an average answer, but description of the diversity of situations, contexts, felt, taken of decision and actions.
  Since this study is observational and descriptive, it does not have a primary judgment criterion, the aim being to describe the studied population. However, according to the method of hierarchical evocation, it can be said that the average frequency of occurrence of the words and their average polarity index will be some outcome measure.

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Cabinet de médecine générale, Beynost
  - Cabinet de médecine générale, Crémieu
  - Cabinet de médecine générale, Lyon
  - Cabinet de médecine générale, Vallon-Pont-d'Arc
  - Cabinet de médecine générale, Vaugneray

IPD SHARING:
Plan to Share IPD: No